CLINICAL TRIAL: NCT07390162
Title: The Effect of Changes in the Frequency of Endotracheal Tube Repositioning in Intensive Care Units on the Prevention of Oral Mucosal Pressure Injuries
Acronym: PreventionMMPI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ecem Ozdemir, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2025/07-02 (KA-24086)-D-Number; 2025/07-02 (KA-24086)-D-Number (Registry Identifier: Turkish Medicines and Medical Devices Agency Ministry of Health of the Republic of Turkey); Clinical Research Ethics C. (Other: Turkish Medicines and Medical Devices Agency Ministry of Health of the Republic of Turkey & Hacettepe University)
Record Dates: First submitted 2025-07-31; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Mucosal Wound; Mucosal Erosion; Mucosal Irritation; Endotracheal Intubation Fixation; Endotracheal Tube Position; Repositioning; Intensive Care Units (ICUs); Adult Patients; Pressure Ulcer Prevention
Keywords: mucosal membrane pressure injury; Intensive Care Units (ICUs); Endotracheal intubation fixation; Repositioning; pressure ulcer prevention

STUDY DESIGN:
Intervention Model Description: Randomization in the study will be performed using Random Allocation Software 2.0, and patients will be randomized into two groups (4 hours and 8 hours) based on the duration of ETT repositioning.
  Inclusion Criteria:
  * Over 18 years of age,
  * Receiving MV support with an oral ETT,
  * No tissue loss/damage in the oral mucosa at the time of admission to the ICU,
  * Less than 24 hours since intubation,
  * APACHE II score ≤24,
  * Patients whose first-degree relatives have given consent for participation in the study will be included.
  Exclusion Criteria:
  * Receiving noninvasive MV support (CPAP-Continuous Positive Airway Pressure/BPAP-Bilevel Positive Airway Pressure),
  * Oncology patients (patients undergoing chemotherapy) will be excluded from the study.
  In the study, patients will be stratified according to their APACHE II scores (APACHE <20---APACHE 20-24).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APACHE II score ≤20 Patients (Experimental)
  Interventions: Other: Changes in the frequency of endotracheal tube repositioning
- APACHE II score 20-24 Patients (Experimental)
  Interventions: Other: Changes in the frequency of endotracheal tube repositioning

INTERVENTIONS:
Other: Changes in the frequency of endotracheal tube repositioning — Ensuring changes in the frequency of endotracheal tube repositioning (two experimental groups of 4 and 8 hours)

SUMMARY:
Intensive care units (ICUs) are care centers equipped with a wide range of technological tools and devices used to provide the highest level of care to individuals whose lives are at risk, requiring a multidisciplinary team approach. Patients may require respiratory support from a ventilator to maintain breathing. In the intensive care unit, patients' breathing is maintained using a medical device called an endotracheal tube (ETT). ETTs can cause injuries due to the constant pressure they exert on the patient's mouth and lip area. Therefore, nurses must secure the ETT at specific times to different points in the mouth area (right and left sides of the mouth) to prevent these injuries. Injuries to the mucosa caused by medical equipment are defined as "mucosal membrane pressure injuries (MMPI)." One such injury is an injury to the mouth. Injuries occurring in the mouth are caused by the pressure of the tubes that enable the patient to breathe in and out.

"The Effect of Changes in the Frequency of Endotracheal Tube Repositioning in Intensive Care Units on the Prevention of Oral Mucosal Pressure Injuries" is a doctoral thesis study; the aim of this study is to investigate the effect of differences in the time interval for changing the position of the tube in the lip region on the prevention of injuries occurring in the mouth in patients monitored with ETT in the ICU. A review of the literature revealed that there are gaps in studies conducted at the international or national level on this subject, and that there is no definitive time guideline for changing (repositioning) the tube in the lip area.

The study will include patients over the age of 18 who are being monitored with an ETT in their mouth, who did not have any injuries in the mouth area at the time of admission to the ICU, who have not had the tube in their mouth for more than 24 hours, who are in moderate to good general condition, and whose first-degree relatives have given permission for them to participate in the study. In the study, the follow-up and evaluation of patients will be limited to six days after tube insertion. Patients who do not require respiratory support with ETT and oncology patients (patients undergoing chemotherapy) will be excluded from the study. Patients who are discharged or transferred during the seven-day follow-up period will be excluded from the study. According to the sample calculation for the study, a total of 230 patients (115 volunteers in the 4-hour group and 115 volunteers in the 8-hour group) will be sufficient. ICU nurses are not bound by any specific time for securing the ETT. Nurses positioned the tube fixation site at the right lip edge/left lip edge/mid-lip line; however, since they were not bound by a specific time-based rule, tube care was nurse-specific. In this study, the location of tube fixation will be recorded through observation to determine the effect of tube fixation on the formation of oral injuries. This study is planned to be completed within a 24-month timeframe between June 15, 2025, and June 15, 2027.

This research is a scientific research (doctoral thesis) study. The daily tube care of volunteers is already in place, and we emphasize that this research will not affect/interfere with the treatment and follow-up of volunteers, and that volunteers will not be negatively affected by the study in any way. The principal investigator will randomly assign volunteers being monitored with ETT to groups using a computer system and will request nurses to reposition their ETTs based on the time intervals (4 hours-8 hours) within these groups. At the same time, the researcher will collect relevant clinical data that may affect pressure injuries in patients (age, gender, smoking history, body mass index, medical history, ICU admission diagnosis, SOFA and APACHE II scores, Glasgow Coma Scale, laboratory findings (C-reactive protein, white blood cell, Hemoglobin, Hematocrit, Total Protein, Albumin), Nutritional Status (Route and Type of Nutrition), Medication Support (Sedatives, Inotropes, Antibiotics, Steroids), ETT-Related Data (Number, Depth, Fixation Site, Repositioning Time), Eilers Oral Assessment Guide and Oral Care Frequency, Braden Pressure Ulcer Risk Assessment Scale and Overall Body Pressure Ulcer Presence, Reaper Oral Mucosa Pressure Injury Scale Grade data, etc.). The follow-up period in the study will be seven days, during which the principal investigator will record the patients' personal health data mentioned above and terminate the follow-up of patients who develop pressure injuries in the oral mucosa. Our expectation from the study is that no injuries will occur in the mouth. In the event of a possible injury, the intervention will be terminated immediately.

DETAILED DESCRIPTION:
In the study, the legal representative of the volunteer will be informed in such a case, and the routine tube repositioning schedule (twice a day, every 12 hours) of the intensive care unit will be resumed. The study is being conducted to shorten the frequency of tube repositioning and to prevent oral mucosal pressure injuries. In accordance with Law No. 6698 on the Protection of Personal Data, the volunteers' names, surnames, and Turkish ID numbers will not be collected. Only personal health data related to chronic diseases, age, and the aforementioned pressure injuries, as listed in the data collection form, will be collected by the responsible researcher. Even when the research is published, the volunteers' identity information will remain confidential. The data in the research will be accessible to the ethics committee, the institution, and other relevant health authorities, who will be able to directly access the volunteer's original medical records. However, this information will be kept confidential in accordance with Law No. 6698, and the legal representative will have given permission for such access by signing the written informed consent form. If new information related to the research topic is obtained that could affect the volunteer's desire to continue participating in the research, the legal representative will be informed in a timely manner. The records obtained will be kept by the researchers for a certain period of time and destroyed after 15 years. Participation in this study is entirely voluntary. Volunteers are currently patients receiving treatment in the intensive care unit and have no responsibility for the study. The legal representatives of volunteers are responsible for not disclosing information about the study to outsiders. You have the right to refuse to participate in the study or to withdraw from it at any time after participating. By filling in and signing the box below with your name, you indicate your consent to participate in the study. The information obtained from this study will be used solely for research purposes. You will not be paid for participating in the study.

I have read all the explanations in the Informed Consent Form. The researchers listed below have provided me with written and verbal explanations regarding the research described above. I understand that I am participating in the research voluntarily and that I may withdraw from the research at any time, with or without cause. I agree to participate in the research of my own free will, without any pressure or coercion.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients over the age of 18, receiving MV support with oral ETT, with no tissue loss/damage in the oral mucosa at the time of admission to the ICU, who have been intubated for less than 24 hours, with an APACHE II score ≤24, and whose first-degree relatives have given consent for their participation in the study.

Exclusion Criteria:

* Oncology patients (patients undergoing chemotherapy) receiving MV support with noninvasive methods (CPAP-Continuous Positive Airway Pressure/BPAP-Bilevel Positive Airway Pressure) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Oral mucosal pressure injury formation | The first 7 days of monitoring
  Oral mucosal pressure injury formation was accepted as the primary outcome variable in the study.

IPD SHARING:
Plan to Share IPD: No
Since this is a planned doctoral thesis in the field of nursing, it should remain as it is for now.

REFERENCES:
- [Result] Ozdemir E, Kavakli O. Risk factors for oral mucosal pressure injury associated with endotracheal tubes in intensive care unit patients: A single-centre longitudinal study with brief follow-up. Nurs Crit Care. 2025 Mar;30(2):e70009. doi: 10.1111/nicc.70009. PMID 40068960